CLINICAL TRIAL: NCT02596984
Title: Evaluation of the Pharmacokinetics of Caspofungin in ICU Patients
Acronym: CaspoKin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308173; 140413A-41 (Other: ANSM); 2014-000789-22 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Shock
Keywords: Intensive Care Unit; Shock; Antifungal agent; Pharmacokinetics; Sepsis
MeSH Terms: conditions — Shock; Sepsis | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- caspofungin (Experimental): Caspofungin will be administered according to the international recommendation.
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Either preemptive, empirical or curative prescription of Caspofungin by one of the ICUs' attending physician. Caspofungin will be administered according to the international recommendation

SUMMARY:
Although the pharmacokinetics of Caspofungin has been studied in healthy subjects and patients, only a few studies have been performed in critically-ill patients. In these patients several factors, including sepsis, shock, increased distribution volume, hepatic dysfunction and hypoalbuminemia may result in dramatic changes in antibiotic concentrations and pharmacokinetics. Caspofungin pharmacokinetic data is scarce and are results mainly from case series or animal studies. Thus, studies performed so far show Caspofungin trough concentrations either decreased, similar to usual value in non-critically ill patients or increased. One of these studies suggested that body weight and hypoalbuminemia may be the main factors associated with Caspofungin pharmacokinetic variability. Pharmacokinetic parameters of caspofungin in pigs with hypovolemic shock suggested the peripheral volume of distribution of caspofungin and intercompartmental clearance to be higher than in healthy animals. These results are however preliminary and cannot be extrapolated suggesting further clinical studies in human to be needed.

The primary objective of this study is to assess Caspofungin trough concentrations and pharmacokinetics in critically-ill patients requiring vasopressors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 y.o)
* Either preemptive, empirical or curative prescription of Caspofungin by one of the ICUs' attending physician
* Requiring vasopressors
* Admission in one of the participating ICUs.

Exclusion Criteria:

* Pregnancy
* Lack of affiliation to the National Medical Insurance
* Previous inclusion in the study
* Inclusion in a concomitant study that may interact with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Caspofungin pharmacokinetic : clearance (ml.min-1) | day 2 - day 3 - day 4
Caspofungin pharmacokinetic : volume of distribution (mL) | day 2 - day 3 - day 4

SECONDARY OUTCOMES:
Caspofungin trough concentration | day 2 - day 3 - day 4
proportion of patients for whom the trough concentrations are lower than the MIC (Minimum Inhibitory Concentration) 90 of Candida ( 1mg / L) | day 2 - day 3 - day 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael DARMON, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand
  - Hôpital Saint-Louis, Paris
  - CHU de SAINT-ETIENNE, Saint-Etienne